CLINICAL TRIAL: NCT06398054
Title: Comparison of the Analgesic Efficacy of Ibuprofen Alone and Ibuprofen Plus Hyoscine-n- Butyl Bromide in Reducing Pain of Outpatient Hysteroscopy: a Randomized, Phase iv, Double-blind Trial
Brief Title: A Study to Investigate the Analgesic Efficacy of Ibuprofen Alone and Ibuprofen Plus Hyoscine-n- Butyl Bromide in Reducing Pain of Outpatient Hysteroscopy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Lorenzo Quirino, Principal Investigator, MD, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYSTPAIN
Record Dates: First submitted 2024-04-10; First posted 2024-05-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: hysteroscopy
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Upon confirmation of eligibility, subjects will be randomly assigned (with a 1:1 allocation as per a computer generated randomization list with the same number of patients in each group) into one of two treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Placebo Comparator): will receive one tablet of ibuprofen 400 mg and two tablets of placebo (similar in size, structure and colour to Hyoscine N-Butil Bromide)
  Interventions: Drug: Ibuprofen 400 mg; Drug: placebo
- Ibuprofen plus HHB (Experimental): will assume one tablet of ibuprofen 400 mg plus two tablets of Hyoscine N-Butil Bromid 10 mg.
  Interventions: Drug: Ibuprofen 400 mg; Drug: Hyoscine N-Butil Bromide

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Ibuprofen 400 mg tablet
Drug: Hyoscine N-Butil Bromide — Hyoscine N-Butil Bromide 10 mg two tablets
  Arms: Ibuprofen plus HHB
Drug: placebo — Two tablets
  Arms: Ibuprofen

SUMMARY:
For outpatient hysteroscopy (OH), it is recommended to take a standard dose of NSAIDs or more hyoscine-n butyl bromide (HBB) an hour prior to the procedure to minimize pain during the first postoperative hour. As there is currently no clear consensus in the literature regarding the best approach to pain management associated with office hysteroscopy procedures. This Phase 4 study is being conducted to evaluate the effectiveness of oral ibuprofen alone and in combination with HBB to determine the most appropriate strategy for improving pain perception in outpatients.

DETAILED DESCRIPTION:
This is a randomized, phase IV, double-blind, placebo-controlled clinical trial.

The subjects will be randomly assigned into one of two treatment arms:

* Group A (Ibuprofen ): will receive one tablet of ibuprofen 400 mg and two tablets of placebo (similar in size, structure and colour to HBB)
* Group B (Ibuprofen plus HHB): will assume one tablet of ibuprofen 400 mg plus two tablets of HHB 10 mg.

The purpose of this study is to evaluate the effectiveness of oral ibuprofen alone and in combination with HBB to determine the most appropriate strategy for improving pain perception in outpatients.

ELIGIBILITY:
Inclusion Criteria:

* female patients older than 18 years who signed informed consent;
* patients who need an office hysteroscopy for their diagnosis or treatment. Those indications included postmenopausal endometrial thickening (over 4 mm), metrorrhagia, sonographic suspicion of endometrial polyps or myomas, Essure device insertion, and endometrial biopsy

Exclusion Criteria:

* women with a possible pregnancy, ongoing vaginal bleeding, lower genital tract infection, gestational trophoblastic disease, asthma, hepatitis, renal failure, lactation, previous cervical surgery, or oversensitivity to one of the agents or their elements;
* patients suffering from neuropathic pain or other conditions that can impact on the perception of pain;
* individuals who use antidepressant, anxiolytics or other drugs/supplements that may have an impact on the perception of pain;
* contraindications to the use of ibuprofen and/or Hyoscine N-Butil Bromide .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by visual analog pain score (10-point VAS, where 0 indicates no pain and 10 indicates the worst possible pain) | During office hysteroscopy procedure, 5 minutes after office hysteroscopy procedure, 30 minutes after hysteroscopy procedure
  The primary objective of this study is to determine the effectiveness of the use of ibuprofen 400 mg alone or a combination of 400 mg ibuprofen and 20 mg Hyoscine N-Butil Bromide, one hour before office hysteroscopy, has a different impact on reducing pain in patients.

SECONDARY OUTCOMES:
Visual analog pain score for pain assessment (10-point VAS, where 0 indicates no pain and 10 indicates the worst possible pain) | During office hysteroscopy procedure, 5 minutes after office hysteroscopy procedure, 30 minutes after hysteroscopy procedure
  To assess a different response to analgesic treatment between nullipare and multipare
Use of Visual analog pain score (10-point VAS, where 0 indicates no pain and 10 indicates the worst possible pain) | 5 minutes after office hysteroscopy procedure, 30 minutes after hysteroscopy procedure
  To evaluate response in post menopausal condition
Measure of the level of anxiety (through STAI-Y1 items, with a score from 1 to 4, where: 1 = not at all and 4 = very much) | During office hysteroscopy
  Measure of the level of pre-procedural anxiety through the STAI-Y (scoring range: 20-80; cut-off: 39-40)
Rate of adverse effects (percentage of events collected) | up to 24 hours
  Determine the safety profile of the study medications

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Quirino, Principal Investigator — ASST Fatebenefratelli Sacco

IPD SHARING:
Plan to Share IPD: No